CLINICAL TRIAL: NCT04698174
Title: Prospective Clinical Study to Evaluate the Safety and Efficacy of a New Transepithelial Photorefractive Keratectomy Treatment
Brief Title: Safety and Efficacy of a New Transepithelial Photorefractive Keratectomy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BL1902
Record Dates: First submitted 2020-10-30; First posted 2021-01-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-03

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transepithelial Photorefractive keratectomy (tPRK) without laser polishing (Experimental)
  Interventions: Procedure: Transepithelial Photorefractive keratectomy (tPRK) without laser polishing
- Transepithelial Photorefractive keratectomy (tPRK) with laser polishing (Experimental)
  Interventions: Procedure: Transepithelial Photorefractive keratectomy (tPRK) with laser polishing
- Standard Photorefractive keratectomy (PRK) (Active Comparator)
  Interventions: Procedure: Standard Photorefractive keratectomy (PRK)

INTERVENTIONS:
Procedure: Transepithelial Photorefractive keratectomy (tPRK) without laser polishing — Transepithelial Photorefractive keratectomy (tPRK) with laser ablation of the corneal epithelium and stroma in a single-step procedure using the B+L Teneo 317 Model 2 Excimer Laser.
  Arms: Transepithelial Photorefractive keratectomy (tPRK) without laser polishing
Procedure: Transepithelial Photorefractive keratectomy (tPRK) with laser polishing — Transepithelial Photorefractive keratectomy (tPRK) using the B+L Teneo 317 Model 2 Excimer Laser with end-treatment laser polishing using a fixed thickness of the additional layer of 5 μm.
  Arms: Transepithelial Photorefractive keratectomy (tPRK) with laser polishing
Procedure: Standard Photorefractive keratectomy (PRK) — Conventional Photorefractive keratectomy (PRK) with alcohol-assisted epithelium ablation. Then the aspheric ablation profile will be performed using the B+L Teneo 317 Model 2 Excimer Laser.
  Arms: Standard Photorefractive keratectomy (PRK)

SUMMARY:
This is a prospective, comparative, randomized, controlled, single-blind, single-surgeon, single-center PMCF clinical study whereby participants undergoing refractive surgery for correction of ametropia will receive a transepithelial PRK (tPRK) and conventional PRK treatment in the contralateral eye. To avoid bias in the clinical outcomes, the two PRK treatment options are randomized to the eyes of the patients based on ocular dominance. In addition, a 1:1 randomization is applied within the tPRK group to eyes with and without end-treatment laser polishing.

Both procedures, standard PRK and tPRK, are performed in a one-step procedure. The main difference between the procedures is, that in conventional PRK, the epithelium will be removed using alcohol, whereas in tPRK procedures, the epithelium will be removed by laser ablation.

ELIGIBILITY:
Inclusion Criteria:

* Ametropia
* Myopic subjects with refractive spherical equivalent (MRSE) between -1.5D and -9.0D
* Hyperopic subjects with refractive spherical equivalent (MRSE) between +1.5D and +5.25D
* Signed informed consent form

Exclusion Criteria:

* Ocular comorbidity
* Subject taking systemic medications likely to affect wound healing such as corticosteroids or antimetabolites.
* Subjects who are known to be pregnant, lactating, or who plans to become pregnant over the medications used for standard tPRK.
* Subjects participating in any other ophthalmic clinical trial during this clinical study.
* Subjects with cognitive impairments or other vulnerable persons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Absolute refractive predictability | 3 months follow up
  Absolute refractive predictability is the absolute difference between intended and achieved Manifest Refraction Spherical Equivalent (MRSE) between eyes

SECONDARY OUTCOMES:
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions.
Monocular Uncorrected Distance Visual Acuity (UDVA) under mesopic light conditions | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under mesopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions. Corrected means spectacle corrected.
Monocular Corrected Distance Visual Acuity (CDVA) under mesopic light conditions | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under mesopic light conditions. Corrected means spectacle corrected.
Monocular Contrast Sensitivity | 3 months follow up
  The contrast sensitivity test consists in assessing the possibility to distinguish the alternation of white and grey fringes of difference contrast with difference frequency.
  Contrast sensitivity will be assessed under photopic and mesopic light conditions using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) device at 2.5 m.
Halo Photic phenomena | 3 months follow up
  The amount and disturbance of photic halo side effects will be assessed by the Halo Simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of halo. The simulator utilizes a numerical scale to quantify the size and intensity of halos, ranging from 0 (none), 25 (mild), 50 (moderate), 75 (severe) to 100 (very severe).
Glare Photic phenomena | 3 months follow up
  The amount and disturbance of photic glare side effects will be assessed by the Glare simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of glare. The simulator utilizes a numerical scale to quantify the size and intensity of glare, ranging from 0 (none), 25 (mild), 50 (moderate), 75 (severe) to 100 (very severe).
Corneal pain | 3 months follow up
  The epithelial healing process after photorefractive keratectomy treatment often comes along with the perception of some corneal pain. To assess the pain level, the participants will receive a self-administered pain questionnaire to fill out every day from the day of the surgery until they return for the 6-9 days follow up visit. An 11-point scale will be used to rate the self-reporting of pain, where 0 is 'None' and 10 is the highest level of 'Severe'. Higher scores indicate higher level of pain.
Visual perception scale | 3 months follow up
  To assess the visual perception level, the participants will receive a self-administered visual perception questionnaire to fill out every day from the day of the surgery until they return for the 6-9 days follow up visit. A 4-point scale will be used to rate the self-reporting of visual perception, with 1 = 'Clear' and 4 = 'Very Poor' vision. Higher scores indicate poorer visual perception.

OTHER OUTCOMES:
Absolute refractive predictability | 6 months follow up
  Absolute refractive predictability is the absolute difference between intended and achieved Manifest Refraction Spherical Equivalent (MRSE) between eyes
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 6 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions.
Monocular Uncorrected Distance Visual Acuity (UDVA) under mesopic light conditions | 6 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under mesopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 6 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m, 80 cm and 40 cm in LogMAR scale under photopic light conditions. Corrected means spectacle corrected.
Monocular Corrected Distance Visual Acuity (CDVA) under mesopic light conditions | 6 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m, 80 cm and 40 cm in LogMAR scale under mesopic light conditions. Corrected means spectacle corrected.
Halo Photic phenomena | 6 months follow up
  The amount and disturbance of photic halo side effects will be assessed by the Halo Simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of halo. The simulator utilizes a numerical scale to quantify the size and intensity of halos, ranging from 0 (none), 25 (mild), 50 (moderate), 75 (severe) to 100 (very severe).
Glare Photic phenomena | 6 months follow up
  The amount and disturbance of photic glare side effects will be assessed by the Glare simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of glare. The simulator utilizes a numerical scale to quantify the size and intensity of glare, ranging from 0 (none), 25 (mild), 50 (moderate), 75 (severe) to 100 (very severe).
Corneal pain | 6 months follow up
  The epithelial healing process after photorefractive keratectomy treatment often comes along with the perception of some corneal pain. To assess the pain level, the participants will receive a self-administered pain questionnaire to fill out every day from the day of the surgery until they return for the 6-9 days follow up visit. An 11-point scale will be used to rate the self-reporting of pain. Higher scores indicate higher level of pain, where 0 is 'None' and 10 is the highest level of 'Severe'. Higher scores indicate higher level of pain.
Visual perception scale | 6 months follow up
  To assess the visual perception level, the participants will receive a self-administered visual perception questionnaire to fill out every day from the day of the surgery until they return for the 6-9 days follow up visit. A 4-point scale will be used to rate the self-reporting of visual perception, with 1 = 'Clear' and 4 = 'Very Poor' vision. Higher scores indicate poorer visual perception.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ang, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ang RET. Transepithelial Versus Conventional PRK: A Randomized Controlled Study. Ophthalmol Ther. 2025 Jul;14(7):1567-1579. doi: 10.1007/s40123-025-01167-2. Epub 2025 May 30. PMID 40445504